CLINICAL TRIAL: NCT03455530
Title: Work Should Not Hurt You: Reduction of Hazardous Exposures in Small Businesses Through a Community Health Worker Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Sonora Environmental Research Institute, Inc. (Unknown); El Rio Community Health Center (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: R01ES028250 (NIH); R01ES028250 (NIH)
Record Dates: First submitted 2018-02-21; First posted 2018-03-06 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-03

CONDITIONS: Community Health Aides; Industrial Hygiene; Volatile Organic Compounds

STUDY DESIGN:
Intervention Model Description: Both groups will receive a baseline exposure assessment and health screenings from El Rio Community Health Center. Then, the intervention group will receive the industrial hygiene (IH)-enhanced community health worker (CHW) intervention. After the second exposure assessment, the delayed group will receive the intervention. A third exposure assessment will be obtained to determine if exposure levels and controls are maintained in the intervention group, and to assess the intervention in the delayed group. This will help us assess sustainability of the intervention. CHWs will accompany evaluators during the first assessment but leave before data collection begins. We anticipate that the CHW intervention will be completed over a 60-day time period (range: 30-90 days).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data collection will be conducted by research staff blinded to the intervention condition. CHWs will only be present at the first baseline-assessment prior to data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive the IH-enhanced CHW intervention before (~3 months) the other arm (Delayed Intervention Group).
  Interventions: Other: Industrial Hygiene-Enhance Community Health Worker Intervention
- Delayed Intervention Group (Other): The delayed intervention group will receive the IH-enhanced CHW intervention after (~3 months) the other arm (Intervention Group).
  Interventions: Other: Industrial Hygiene-Enhance Community Health Worker Intervention

INTERVENTIONS:
Other: Industrial Hygiene-Enhance Community Health Worker Intervention — The intervention will be derived from audits and exposure assessments and focus groups with workers and owners in the same business types (excluded from the trial) conducted in an earlier part of the study, as well as a community advisory group (e.g., Hispanic Chamber of Commerce) . From this, we will generate educational materials specific for each small business sector. We will provide the CHWs with a list of industry-specific control options along with potential cost savings and benefits. For example, EPA estimates a cost saving of $13,000 per year for auto body shops that switch to the high-velocity low-pressure spray guns. Each list will be a comprehensive menu of options that contain multiple control measures including simple controls, such as keeping the lids on the solvent containers.

SUMMARY:
This project aims to reduce negative health outcomes in small businesses that primarily employ high-risk Latino workers by characterizing their exposures to hazardous chemicals and assessing if a community health worker (CHW) intervention is effective at decreasing these exposures. Although preventable by definition, occupational disease and injuries are leading causes of death in the United States, with a disproportionate burden faced by Latinos. Small businesses pose a particular risk. They are more likely to employ low-wage Latino workers, and often use hazardous solvents including volatile organic chemicals that can cause asthma, cancer, cardiovascular, and neurological disease; yet their workers lack access to culturally and linguistically appropriate occupational health and pollution prevention information due to economic, physical, and social barriers. CHW-led interventions and outreach in Latino communities have documented increased access to health care and health education and reduced workplace exposures among farmworkers. CHWs are an innovative method to bridge the gap between these small business communities and other stakeholders. The proposed project will capitalize on established partnerships between the University of Arizona, the Sonora Environmental Research Institute, Inc. and the El Rio Community Health Center. A community-engaged research framework will be used to complete the following specific aims: 1) quantify and identify exposures to hazardous chemicals in the two high risk small business sectors common in our target area (i.e., auto repair shops and beauty salons); 2) work collaboratively with business owners, trade groups, workers and CHWs to design an industrial hygiene - enhanced CHW intervention tailored for each small business sector; and 3) conduct a cluster randomized trial to evaluate the effectiveness of the CHW intervention at reducing workplace exposures to volatile organic compounds and assess which factors led to successful utilization of exposure control strategies in both male and female-dominated businesses. Businesses will be randomized to either an intervention or delayed intervention group, both of which will receive incentives to participate including worksite health screenings. CHWs will work closely with business owners and employees to select and implement exposure-strategies appropriate for their worksite using a menu of complementary strategies of varying complexity and cost. This innovative project has the potential to directly reduce occupational health disparities through a CHW intervention that moves beyond providing occupational health education. The intervention will overcome current barriers by helping marginalized Latino workers and small business owners who may have limited education, literacy, and computer skills to understand the hazards associated with their work, and will empower them to have greater control over their occupational exposures, with the ultimate goal of preventing occupational disease and reducing health disparities.

ELIGIBILITY:
Inclusion Criteria:

* workers or owners of small businesses in select sectors (e.g., beauty salons, auto shops) in target zip codes in southern metropolitan Tucson, Arizona

Exclusion Criteria:

* age less than 18 years or people not employed in targeted sectors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sonora Environmental Research Institute, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Result] Davidson KW, Goldstein M, Kaplan RM, Kaufmann PG, Knatterud GL, Orleans CT, Spring B, Trudeau KJ, Whitlock EP. Evidence-based behavioral medicine: what is it and how do we achieve it? Ann Behav Med. 2003 Dec;26(3):161-71. doi: 10.1207/S15324796ABM2603_01. PMID 14644692
- [Result] Kraemer HC, Kuchler T, Spiegel D. Use and misuse of the consolidated standards of reporting trials (CONSORT) guidelines to assess research findings: comment on Coyne, Stefanek, and Palmer (2007). Psychol Bull. 2009 Mar;135(2):173-8; discussion 179-82. doi: 10.1037/0033-2909.135.2.173. PMID 19254073
- [Result] Campbell MK, Elbourne DR, Altman DG; CONSORT group. CONSORT statement: extension to cluster randomised trials. BMJ. 2004 Mar 20;328(7441):702-8. doi: 10.1136/bmj.328.7441.702. No abstract available. PMID 15031246

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Business
Groups:
- Intervention Group - Beauty Salon; Intervention Group - Auto Shops: The intervention group will receive the IH-enhanced CHW intervention before (~3 months) the other arm (Delayed Intervention Group).
  Industrial Hygiene-Enhance Community Health Worker Intervention: The intervention will be derived from audits and exposure assessments and focus groups with workers and owners in the same business types (excluded from the trial) conducted in an earlier part of the study, as well as a community advisory group (e.g., Hispanic Chamber of Commerce) . From this, we will generate educational materials specific for each small business sector. We will provide the CHWs with a list of industry-specific control options along with potential cost savings and benefits. For example, EPA estimates a cost saving of $13,000 per year for auto body shops that switch to the high-velocity low-pressure spray guns. Each list will be a comprehensive menu of options that contain multiple control measures including simple controls, such as keeping the lids on the solvent containers.
- Delayed Intervention Group - Beauty Salon; Delayed Intervention - Auto Shops: The delayed intervention group will receive the IH-enhanced CHW intervention after (~3 months) the other arm (Intervention Group).
  Industrial Hygiene-Enhance Community Health Worker Intervention: The intervention will be derived from audits and exposure assessments and focus groups with workers and owners in the same business types (excluded from the trial) conducted in an earlier part of the study, as well as a community advisory group (e.g., Hispanic Chamber of Commerce) . From this, we will generate educational materials specific for each small business sector. We will provide the CHWs with a list of industry-specific control options along with potential cost savings and benefits. For example, EPA estimates a cost saving of $13,000 per year for auto body shops that switch to the high-velocity low-pressure spray guns. Each list will be a comprehensive menu of options that contain multiple control measures including simple controls, such as keeping the lids on the solvent containers.
Period: Overall Study
Arm/Group | Intervention Group - Beauty Salon | Delayed Intervention Group - Beauty Salon | Intervention Group - Auto Shops | Delayed Intervention - Auto Shops
Started | 77; 23 Business | 70; 23 Business | 69; 19 Business | 52; 19 Business
Completed | 68; 19 Business | 69; 22 Business | 66; 17 Business | 49; 17 Business
Not Completed | 9; 4 Business | 1; 1 Business | 3; 2 Business | 3; 2 Business
Not completed — Withdrawal by Subject | 9 | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Population: This is a cluster-randomized trial where the clusters were businesses. 1-4 workers participated per business.
Groups:
- Intervention Group - Auto Shop: The intervention group will receive the IH-enhanced CHW intervention before (~3 months) the other arm (Delayed Intervention Group).
  Industrial Hygiene-Enhance Community Health Worker Intervention: The intervention will be derived from audits and exposure assessments and focus groups with workers and owners in the same business types (excluded from the trial) conducted in an earlier part of the study, as well as a community advisory group (e.g., Hispanic Chamber of Commerce) . From this, we will generate educational materials specific for each small business sector. We will provide the CHWs with a list of industry-specific control options along with potential cost savings and benefits. For example, EPA estimates a cost saving of $13,000 per year for auto body shops that switch to the high-velocity low-pressure spray guns. Each list will be a comprehensive menu of options that contain multiple control measures including simple controls, such as keeping the lids on the solvent containers.
- Delayed Intervention Group - Auto Shop: The delayed intervention group will receive the IH-enhanced CHW intervention after (~3 months) the other arm (Intervention Group).
  Industrial Hygiene-Enhance Community Health Worker Intervention: The intervention will be derived from audits and exposure assessments and focus groups with workers and owners in the same business types (excluded from the trial) conducted in an earlier part of the study, as well as a community advisory group (e.g., Hispanic Chamber of Commerce) . From this, we will generate educational materials specific for each small business sector. We will provide the CHWs with a list of industry-specific control options along with potential cost savings and benefits. For example, EPA estimates a cost saving of $13,000 per year for auto body shops that switch to the high-velocity low-pressure spray guns. Each list will be a comprehensive menu of options that contain multiple control measures including simple controls, such as keeping the lids on the solvent containers.
- Total: Total of all reporting groups
Arm/Group | Intervention Group - Beauty Salon | Delayed Intervention Group - Beauty Salon | Intervention Group - Auto Shop | Delayed Intervention Group - Auto Shop | Total
Number analyzed (Participants) | 77 | 70 | 69 | 52 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12) | 47 (14) | 40 (12) | 38 (11) | 42.4 (12.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 7 | 7 | 64 | 48 | 126
  Female | 68 | 62 | 4 | 3 | 137
  Unknown | 2 | 1 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 52 | 47 | 37 | 190
  Not Hispanic or Latino | 21 | 15 | 21 | 14 | 71
  Unknown or Not Reported | 2 | 3 | 1 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 77 | 70 | 69 | 52 | 268

OUTCOME MEASURES:

1. Primary Outcome: Change in Volatile Organic Chemical Concentrations From Pre- to Post-Intervention
Description: The primary outcome is the change in average total volatile organic chemical exposures for each business from pre- to post- intervention.
Time Frame: 6 months
Population: This is a cluster-randomized trial where the clusters were small businesses. There were 1-4 workers at each shop per assessment. The unit of analysis here is the average total volatile organic chemicals exposures for each business at each analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: ppb
Units Other Than Participants: Business
Arm/Group | Intervention Group - Beauty Salon | Delayed Intervention Group - Beauty Salon | Intervention Group - Auto Shops | Delayed Intervention - Auto Shops
Number analyzed (Participants) | 68 | 69 | 66 | 49
Number analyzed (Business) | 19 | 22 | 17 | 17
ppb | 2738 [1720 to 4358] | 3875 [2471 to 6077] | 523 [267 to 1026] | 225 [116 to 435]
Statistical Analysis 1: Comparison: Intervention Group - Beauty Salon vs Delayed Intervention Group - Beauty Salon; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [0.45 to 1.19] — Ratio based on the mean difference from the log scale
Statistical Analysis 2: Comparison: Intervention Group - Auto Shops vs Delayed Intervention - Auto Shops; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 1.34, 95% CI 2-sided [0.55 to 3.24] — Ratio based on the mean difference from the log scale

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Intervention Group - Beauty Salon | Delayed Intervention Group - Beauty Salon | Intervention Group - Auto Shop | Delayed Intervention Group - Auto Shop
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/70 | 0/69 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/70 | 0/69 | 0/52
Other Adverse Events (participants affected / at risk) | 0/77 | 0/70 | 0/69 | 0/52

LIMITATIONS AND CAVEATS:
The analysis was performed by business. Workers may have changed during assessment. We were not able to recruit the initial number of businesses due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT03455530/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03455530/SAP_001.pdf